CLINICAL TRIAL: NCT05372107
Title: A Multicenter, Double-Masked, Phase 1b Study Evaluating the Safety, Tolerability, and Dose-Response of Topical AG-80308 in Patients With Dry Eye Disease
Brief Title: A Study of AG-80308 in Dry Eye Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allgenesis Biotherapeutics Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P1-80308-001
Record Dates: First submitted 2022-05-08; First posted 2022-05-12 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): One drop of 0.001% AG-80308, two times daily to both eyes for 3 months
  Interventions: Drug: AG-80308
- Group 2 (Experimental): One drop of 0.03% AG-80308, two times daily to both eyes for 3 months
  Interventions: Drug: AG-80308
- Group 3 (Experimental): One drop of 0.1% AG-80308, two times daily to both eyes for 3 months
  Interventions: Drug: AG-80308
- Group 4 (Experimental): One drop of 0.03% AG-80308, new formulation, two times daily to both eyes for 3 months
  Interventions: Drug: AG-80308

INTERVENTIONS:
Drug: AG-80308 — AG-80308 Eye Drop Solution
  Other Names: AGN-232411

SUMMARY:
This is a multicenter, double-masked, randomized, parallel-group study with topical AG-80308 eye drops in dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older at the screening visit
2. Diagnosis of dry eye disease in both eyes with or without meibomian gland disease

Exclusion Criteria:

1. Participation in any investigational study within 30 days prior to baseline or exposure to an investigational drug must be fully washed out (at least 5 half-lives)
2. Any ocular infection or inflammation within 30 days prior to the screening visit
3. Corneal disorder or abnormalities other than dry eye disease that impact normal spreading of the tear film (except superficial punctate keratitis)
4. History of chronic ocular allergy, systemic lupus erythematosus, rheumatoid arthritis, corneal ulcer/erosions, uveitis or dry eye due to Stevens Johnson syndrome, irradiation, alkali burns, cicatricial pemphigoid or vitamin A deficiency.
5. Use of contact lenses in either eye within 14 days of screening visit or planned use during the study
6. Use of the dry eye and/or meibomian gland disease medications/procedures within 2 to 8 weeks prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events (AEs) and serious AEs (SAEs) | Screening to 3 months

OTHER OUTCOMES:
Mean change from baseline in ocular surface staining | Screening to 3 months
Mean change from baseline in dry eye symptoms | Screening to 3 months
Mean change from baseline in Schirmer's test | Screening to 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Eye Research Foundation, Newport Beach, California
  - Andover Eye Associates, Raynham, Massachusetts
  - Alpine Research Organization, Inc., Clinton, Utah

IPD SHARING:
Plan to Share IPD: No